CLINICAL TRIAL: NCT01400113
Title: Treating Acutely Agitated Patients With Asenapine Sublingual Tablets: A Single-Dose, Randomized, Double-Blind Placebo Controlled Trial
Brief Title: Treating Acutely Agitated Patients With Asenapine Sublingual Tablets
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Principal Investigator, Michael J. Pratts, M.D., Psychiatrist, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P00184
Record Dates: First submitted 2011-07-18; First posted 2011-07-22 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Agitation
Keywords: Acute Agitation; schizophrenia; bipolar; psychosis; panss-ec
MeSH Terms: conditions — Psychomotor Agitation; Schizophrenia; Psychotic Disorders | interventions — asenapine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asenapine (Experimental): This group received 10mg asenapine sl x 1 dose
  Interventions: Drug: Asenapine
- Placebo (Placebo Comparator): This group received placebo sl x 1 dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Asenapine — Asenapine Sublingual Tablet 10mg, single-dose
  Other Names: Saphris
  Arms: Asenapine
Drug: Placebo — Placebo Sublingual Tablet, single-dose
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Our proposal is to administer asenapine to patients who are clinically agitated and in need of immediate intervention. At present there are no controlled studies that we know of that explores the use of asenapine for this purpose. Establishing the utility of asenapine for this common clinical problem will support its use as an additional treatment option in acutely agitated patients.

DETAILED DESCRIPTION:
A psychiatrist (blinded) will assess the patient for agitation and their capacity to consent. Patients will be informed about the study and asked to complete informed consent prior to being included in the study. Patients who decline will not be included. A nurse (blinded) will administer either 10mg asenapine or placebo sublingually in a randomized fashion. Efficacy in reducing acute agitation will be evaluated using the PANSS-EC. A trained rater (blinded) will rate patients at baseline and at 15, 30, 60, 90 and 120 minutes (or endpoint) after medication administration. Efficacy in reducing acute agitation will also be evaluated using the Clinical Global Impression Scale (CGI). A trained rater (blinded) will rate patients at baseline CGI-Severity and CGI-Change at 60 and 120 minutes (or endpoint) after medication administration. The need for additional medications, interventions or physical restraints will be recorded and constitute the endpoint for that patient. Demographics, diagnoses, blood alcohol level, urine toxicology, and urine pregnancy will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be between the ages of 18 and 65
* Be acutely agitated as determined by a total score of ≧ 14 on the PANSS-EC and at least one individual item score of ≧ 4
* Patients must have the capacity to provide informed consent, and such consent will be obtained prior to participation

Exclusion Criteria:

* Patient is knowingly pregnant
* Patient is less than 18 or greater than 65 years old
* Patient had a past adverse or allergic response to Asenapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pratts, MD, Principal Investigator — St. Joseph's Hospital Health Center - CPEP; Laura Leso, MD, Principal Investigator — St. Joseph's Hospital Health Center - CPEP; David Frey, MD, Principal Investigator — St. Joseph's Hospital Health Center - CPEP
Locations (1):
- St. Joseph's Hospital Health Center-Comprehensive Psychiatric Emergency Program (CPEP), Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All data available upon request.

REFERENCES:
- [Derived] Pratts M, Citrome L, Grant W, Leso L, Opler LA. A single-dose, randomized, double-blind, placebo-controlled trial of sublingual asenapine for acute agitation. Acta Psychiatr Scand. 2014 Jul;130(1):61-8. doi: 10.1111/acps.12262. Epub 2014 Mar 10. PMID 24606117

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 4/23/12 and 12/11/12, adult, non-pregnant patients in a Psychiatric Emergency Room were assessed by a psychiatrist for agitation. Those patients who were willing to participate and signed an informed consent were enrolled.
Groups:
- Asenapine; Placebo: 60 patients were randomized to this group
Period: Overall Study
Arm/Group | Asenapine | Placebo
Started | 60 | 60
Completed | 59 | 59
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine | Placebo | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 60 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.1) | 36.4 (12.4) | 36.4 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 43 | 36 | 79
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale - Excited Component
Description: The primary outcome measure is change in the Positive and Negative Syndrome Scale - Excited Component (PANSS-EC) from baseline to 2 hours after medication administration. The PANSS-EC consists of 5 items: excitement, tension, hostility, uncooperativeness, and poor impulse control. The 5 items from the PANSS-EC are rated from 1 (not present) to 7 (extremely severe); scores range from 5 to 35; mean scores ≥ 20 clinically correspond to severe agitation. This set of items detects differences between drug and placebo when evaluating acute agitation and aggression in psychiatric patients with different psychiatric pathologies.
Time Frame: Change in PANSS-EC score from baseline to 2 hours post drug/placebo administration.
Measure: Mean (95% Confidence Interval); unit: PANSS SCORE
Arm/Group | Asenapine | Placebo
Number analyzed (Participants) | 59 | 59
PANSS SCORE | 7.86 [2.06 to 13.66] | 14.93 [7.69 to 22.17]

2. Secondary Outcome: Clinical Global Impression Scale
Description: Secondary outcome measures will include the Clinical Global Impression -Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I) scales.
Time Frame: 2 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Asenapine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
1. The short observation period of 2 hours.
2. Dependence on spontaneous self reporting of adverse effects.
3. Specific inquiry was not made regarding adverse events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes